CLINICAL TRIAL: NCT04922021
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled, Multi-site, Proof of Concept Trial to Evaluate the Efficacy and Safety of LEO 138559 in Adult Subjects With Moderate to Severe Atopic Dermatitis (AD).
Brief Title: An Evaluation of LEO 138559 in Adults With Moderate to Severe Atopic Dermatitis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0145-1376; 2020-005541-16 (EudraCT Number)
Record Dates: First submitted 2021-06-07; First posted 2021-06-10 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2023-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LEO 138559 (Experimental): Participants will receive injections of LEO 138559 from Week 0 (baseline) to Week 16 (end of treatment).
  Interventions: Drug: LEO 138559
- Placebo (Placebo Comparator): Participants will receive injections of placebo from Week 0 (baseline) to Week 16 (end of treatment).
  Interventions: Drug: LEO 138559 placebo

INTERVENTIONS:
Drug: LEO 138559 — LEO 138559 is an antibody given by injection just under the skin.
  Arms: LEO 138559
Drug: LEO 138559 placebo — LEO 138559 placebo is given by injection just under the skin. LEO 138559 placebo contains the same excipients in the same concentration as LEO 138559, except for the medical ingredient LEO 138559.
  Arms: Placebo

SUMMARY:
This is a clinical study in adult participants with moderate to severe atopic dermatitis (AD).

The purpose of the study is to test a new medicine (LEO 138559) given by injection to see if it works to treat AD and what the side effects are when compared with a placebo injection with no medical ingredient.

The study will last up to 36 weeks for each participant. The study will include a treatment period of 16 weeks, during which the participants will receive the injections, followed by a period of 16 weeks without treatment with the main purpose of continuing safety evaluations. The participants will regularly visit the clinic for tests and the study doctor will evaluate their AD. The participants will also be asked to answer questions about their AD symptoms and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old (both included) at screening.
* Diagnosis of atopic dermatitis (AD) (as defined by the American Academy of Dermatology Consensus Criteria) that has been present for ≥1 year prior to screening.
* Subjects who have a recent history (within 6 months before screening) of inadequate response to treatment with topical medication, or for whom topical treatments are otherwise medically inadvisable.
* Eczema Area and Severity Index (EASI) score ≥12 at screening and ≥16 at baseline.
* Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) score ≥3 at screening and baseline.
* Body surface area (BSA) of AD involvement ≥10% at screening and baseline.
* Worst Daily Pruritus Numeric Rating Scale (NRS, weekly average) of ≥3 points at baseline.

Exclusion Criteria:

* Treatment with systemic immunosuppressive/immunomodulating medication, immunoglobulin/blood products, or phototherapy within 4 weeks or 5 half-lives prior to randomization, whichever is longer.
* Treatment with biologics within 5 half-lives (if known) or 16 weeks prior to randomization, whichever is longer.
* Treatment with topical corticosteroid(s) (TCS), topical calcineurin inhibitor(s) (TCI), topical phosphodiesterase-4 (PDE-4) inhibitor, or other topical prescription treatments within 1 week prior to randomization.
* Treatment with a live (attenuated) vaccine within 12 weeks prior to randomization.
* Clinically significant active chronic or acute infection requiring systemic treatment within 4 weeks prior to randomization that may compromise the safety of the subject.
* Skin infection within 1 week prior to the baseline visit.
* Presence of hepatitis B or C infection at screening.
* History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
* Participant has a positive or indeterminate test for tuberculosis at screening.
* Participant is pregnant or lactating.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (16):
- United States (5):
  - LEO Pharma Investigational Site, Birmingham, Alabama
  - LEO Pharma Investigational Site, Fountain Valley, California
  - LEO Pharma Investigational Site, Los Angeles, California
  - LEO Pharma Investigational Site, Doral, Florida
  - LEO Pharma Investigational Site, Hialeah, Florida
- Canada (3):
  - LEO Pharma Investigational Site, Markham, Ontario
  - LEO Pharma Investigational Site, Mississauga, Ontario
  - LEO Pharma Investigational Site, Peterborough, Ontario
- Germany (4):
  - LEO Pharma Investigational Site, Berlin
  - LEO Pharma Investigational Site, Dresden
  - LEO Pharma Investigational Site, Leipzig
  - LEO Pharma Investigational Site, Lübeck
- Poland (4):
  - LEO Pharma Investigational Site, Krakow
  - LEO Pharma nvestigational Site, Rzeszów
  - LEO Pharma Investigational Site, Warsaw
  - LEO Pharma Investigational Site, Wroclaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LEO 138559 | Placebo
Started | 29 | 29
Completed | 22 | 16
Not Completed | 7 | 13
Not completed — Withdrawal by Subject | 4 | 10
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Multiple reasons | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LEO 138559 | Placebo | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (12.1) | 32.8 (10.2) | 35.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 12 | 13 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 26 | 28 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 25 | 24 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 3 | 3 | 6
  United States | 5 | 3 | 8
  Poland | 16 | 19 | 35
  Germany | 5 | 4 | 9
EASI [Mean (Standard Deviation); unit: units on a scale] — The Eczema Area and Severity Index (EASI) is a validated measure used in clinical trials to evaluate the extent and severity of atopic dermatitis. EASI is a composite score ranging from 0 to 72 with higher scores indicating a more extensive and/or severe condition.
  units on a scale | 26.93 (11.77) | 26.12 (9.80) | 26.53 (10.74)
Baseline disease severity [Count of Participants; unit: Participants] — The Eczema Area and Severity Index (EASI) is a validated measure used in clinical trials to evaluate the extent and severity of atopic dermatitis. EASI is a composite score ranging from 0 to 72 with higher scores indicating a more extensive and/or severe condition.
  EASI score < 21 indicated moderate eczema EASI score ≥ 21 indicated severe eczema
  Participants
    Baseline EASI score <21 | 14 | 13 | 27
    Baseline EASI score ≥21 | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change in EASI Score From Baseline to Week 16
Description: The Eczema Area and Severity Index (EASI) is a validated measure used in clinical trials to evaluate the extent and severity of atopic dermatitis. EASI is a composite score ranging from 0 to 72 with higher scores indicating a more extensive and/or severe condition.
Time Frame: Week 0 to Week 16
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | LEO 138559 | Placebo
Number analyzed (Participants) | 29 | 29
score on a scale | -15.3 (2.64) | -3.5 (2.91)
Statistical Analysis 1: Comparison: LEO 138559 vs Placebo; Test type: Superiority — Two-sided hypotheses were tested based on the pre-specified primary analysis for the primary estimand. The primary estimand used a hypothetical strategy evaluating the treatment difference as if all subjects adhered to the treatment regimen, i.e. they did not discontinue IMP permanently, did not initiate rescue treatment, or did not have more than one missed treatment dose related to COVID-19; p = 0.003, ANCOVA — The type I error rate of the two-sided hypothesis test was controlled at the 5% significance level; ANCOVA model: Change in EASI = Treatment + Region + Baseline EASI. Missing values and data 'treated as missing' were imputed using MI assuming MAR; Mean Difference (Net) = -11.8, 95% CI 2-sided [-19.6 to -4.1] — Estimates of difference in LS-means and associated standard errors from the analyses were combined using Rubin's rule to provide the overall pooled estimate and associated standard error. LS-means was estimated using the observed margins for the FAS

2. Secondary Outcome: Number of Treatment-emergent Adverse Events From Baseline to Week 16 Per Subject
Time Frame: Week 0 to Week 16
Measure: Number; unit: adverse events
Arm/Group | LEO 138559 | Placebo
Number analyzed (Participants) | 29 | 29
adverse events | 40 | 26

ADVERSE EVENTS:
Time Frame: 32 weeks (Treatment period: Week 0 to Week 16; Safety follow-up period: Week 16 to Week 32)
Groups:
- LEO 138559: LEO 138559 (N=29)
- Placebo: Placebo (N=29)
Arm/Group | LEO 138559 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 21/29 | 14/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEO 138559 (N=29) | Placebo (N=29)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 1 (1) | 2 (3)
Inflammation (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (3) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 6 (6) | 2 (2)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Eczema herpeticum (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 5 (6)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 (5) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma seeks publication of all Phase 3 clinical trials in peer-reviewed journals within 18 months of trial completion, regardless of whether the findings are positive or negative. If there is no multi-centre publication within 18 months after the clinical trial has been completed or terminated at all trial sites, the investigator has the right to publish the results from the clinical trial generated by the investigator.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-31): https://cdn.clinicaltrials.gov/large-docs/21/NCT04922021/Prot_SAP_000.pdf